CLINICAL TRIAL: NCT02086955
Title: Outpatient Nurse Managed Counseling Program for Patients With Diabetic Foot Ulceration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zurich University of Applied Sciences (Other)
Collaborators: Swiss National Science Foundation (Other); Nursing Science Foundation Switzerland (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Lorenz Imhof, Prof. Dr., Zurich University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 320030_143863; 2010-0278/0 (Other: KEK-ZH-NR)
Record Dates: First submitted 2014-03-03; First posted 2014-03-13 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetes; Nursing counseling; Foot ulceration; Outpatient; Advanced Practice Nurse
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Foot Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (No Intervention): All participants receive three specially-developed brochures with information regarding the diabetic foot condition. The brochures containes explanations to a) the cause and warning signs of diabetic foot ulcers, b) the precautions patients can take in their daily life, and c) helpful foot gymnastics to be practiced at home.
- Nursing counseling (Experimental): The participants who are randomized in the intervention group receive standardized education regarding diabetic foot care. The nurse-led outpatient intervention go on for five weeks. During a period of five weeks, the participants are provided with weekly education, skill training, and counseling sessions on foot care.
  Interventions: Behavioral: Nursing counseling

INTERVENTIONS:
Behavioral: Nursing counseling — The participants who are randomized in the intervention group receive standardized education regarding diabetic foot care. The nurse-led outpatient intervention lasts five weeks. During a period of five weeks, the participants are provided with weekly skill training, and counseling sessions on foot care. Each participant receives a foot care kit with essential foot care material and a foot care diary.
  Arms: Nursing counseling

SUMMARY:
The purpose of the study is to evaluate the effectiveness of a nurse led intervention for high risk patients with diabetic foot ulceration and/or amputation.

The effectiveness is defined in two ways 1) as a reduction in complication rates (time till ulceration recurrence, new ulcerations, amputation or reamputation) and 2) as a reduction in hospital readmissions for foot-related complication (one year survival probability: failure = readmission for ulceration recurrence, new ulcerations, amputation or re-amputation).

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is associates with numerous complications. One of these is decreased peripheral circulation impaired sensation leading to the development of foot ulcers that lead to amputations of toes, feet and limbs. These complications not only have devastating effects on the individual in terms of loss of functionality but also impact the patient's ability to carry out and enjoy occupational, recreational and family functioning activities. Furthermore, foot ulcers and associated problems often lead to prolonged hospitalization and loss of productivity. All of these have personal as well as societal economical implications.

This pilot randomized clinical trial (RCT) aims to evaluate the feasibility of an additional patient education program to current management of foot care in patients with DM.

The study aims to test an alternative to current standard of care for patients with foot ulcers. A RCT is the preferred method to establish efficacy for this alternative nurse managed intervention; and if found to be effective, the current study will also allow an evaluation of the cost effectiveness of this intervention and the potential economic reduction in cost to the health care system.

The potential implications are major in terms of quality of life, reduction in morbidity in disability days, and cost savings. It is anticipated that this intervention is at least as effective as hospital stay, and being surrounded by their own loved ones without the threats that a hospital setting presents. The findings will be important to consider whether clinical practice can be changed to benefit patients. If the study results show that the subjects in the IG have better skills in monitoring and treating their diabetic foot ulcerations and eventually avoid developing further complications the intervention can be applied to future patients.

ELIGIBILITY:
Inclusion Criteria:

* patients age 18 or older
* in current treatment for ulceration and/or amputation of a lower limb
* are able to understand German oral and in writing
* are able to give written informed consent

Exclusion Criteria:

* severe psychiatric diagnoses
* subjects living in dependent living facilities (nursing home or rehabilitation)
* subjects lacking supporting family members and incapable of selfmonitoring their feet due to impairment (vision or physical movement)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2013-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of nurse-led intervention for high risk patients with diabetic foot ulceration/amputation | Participants will be followed for the duration of 42 weeks. Data will be collected at baseline (T0) as well as after 5 weeks (T1), 12 weeks (T2), 24 weeks (T3) and after 42 weeks (T4).
  After the baseline data collection (T0), data will be collected after 5 weeks (T1), 12 weeks (T2), 24 weeks (T3) and after 42 weeks (T4) regarding:
  - foot related complications (hospital readmission for ulceration recurrence, new ulcerations or amputations)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz Imhof, Prof. Dr., Principal Investigator — University of applied sciences
Locations (1):
- Zurich University of Applied Sciences, Winterthur, Canton of Zurich, Switzerland